CLINICAL TRIAL: NCT05780424
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With COVID-19 (Trial H3: BRII-196/BRII-198)
Brief Title: BRII-196/BRII-198 for Inpatients With COVID-19 (An ACTIV-3/TICO Treatment Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (Other); Cardiothoracic Surgical Trials Network (Other); Brii Biosciences Limited (Industry); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 014/ACTIV-3/H3
Record Dates: First submitted 2023-03-20; First posted 2023-03-22 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Infections; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3; TICO
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — amubarvimab; romlusevimab; remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BRII-196/BRII-198 plus SOC (Experimental): * BRII-196 1000 mg solution; administered as IV infusion
  * BRII-198 1000 mg solution; administered as IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Biological: BRII-196; Biological: BRII-198; Biological: Remdesivir
- Placebo plus SOC (Placebo Comparator): * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Biological: Placebo; Biological: Remdesivir

INTERVENTIONS:
Biological: BRII-196 — BRII-196 is a fully human immunoglobulin G (IgG)-1 monoclonal antibody (mAb) derived from antibody P2C-1F11 that was isolated directly from human B cells of a convalescent COVID-19 patient.
  Arms: BRII-196/BRII-198 plus SOC
Biological: BRII-198 — BRII-198 is a fully human IgG-1 mAb derived from antibody P2B-1G5 that was isolated directly from human B cells of a convalescent COVID-19 patient.
  Arms: BRII-196/BRII-198 plus SOC
Biological: Placebo — Commercially available 0.9% sodium chloride solution
  Arms: Placebo plus SOC
Biological: Remdesivir — Antiviral agent
  Other Names: Veklury

SUMMARY:
This study looks at the safety and effectiveness of BRII-196/BRII-198 in treating COVID-19 in people who have been hospitalized with the infection. Participants in the study will be treated with either BRII-196/BRII-198 plus current standard of care (SOC), or with placebo plus current SOC. This is ACTIV-3/TICO Treatment Trial H3.

DETAILED DESCRIPTION:
This is a treatment trial of the ACTIV-3/TICO master protocol (NCT04501978) to evaluate the safety and efficacy of BRII-196/BRII-198 in hospitalized patients infected with COVID-19.

This is a randomized, blinded, controlled sub-study of BRII-196/BRII-198 plus current standard of care (SOC) against placebo plus current SOC. The placebo arm may be shared across other sub-studies of the ACTIV-3/TICO master protocol. When more than one drug is being tested at the same time, participants will be randomly allocated to treatments or placebo.

Randomization will be stratified by study site pharmacy and disease severity. There are 2 disease severity strata: Participants without organ failure (severity stratum 1) and participants with organ failure (severity stratum 2).

An independent Data and Safety Monitoring Board (DSMB) will regularly review interim analyses and summarize safety and efficacy outcomes. The pace of enrollment with be initially restricted, and there will be an early review of safety data by the DSMB. At the outset of the trial, only participants in disease severity stratum 1 will be enrolled. This will continue until approximately 300 participants are enrolled and followed for 5 days. The exact number will vary according to the speed of enrollment and the timing of DSMB meetings. Prior to expanding enrollment to also include patients in disease severity stratum 2, safety will be evaluated and a pre-specified futility assessment by the DSMB will be carried out using 2 ordinal outcomes assessed at Day 5.

If BRII-196/BRII-198 passes the futility assessment, enrollment of participants will be expanded, seamlessly and without any data unblinding, to include participants in disease severity stratum 2 as well as those in disease severity stratum 1. Future interim analyses will be based on the primary endpoint of sustained recovery and will use pre-specified guidelines to determine early evidence of benefit, harm, or futility for the investigational agent. Participants will be followed for 18 months following randomization.

This trial will be conducted in several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

ELIGIBILITY:
Inclusion Criteria:

* Refer to the master protocol (NCT04501978)

Exclusion Criteria:

* Refer to the master protocol (NCT04501978)
* Additional Exclusion Criteria:

  * Pregnant women
  * Nursing mothers
* In addition, prior to the initial futility assessment which is performed when approximately 150 participants have been enrolled on BRII-196/BRII-198 and 150 on placebo, patients on high-flow oxygen or non-invasive ventilation (category 5 of the pulmonary ordinal outcome) will be excluded. These patients may be eligible for the trial if the initial futility assessment is passed by this agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lundgren, Prof., Principal Investigator — INSIGHT Copenhagen International Coordinating Centre, Rigshospitalet, University of Copenhagen; James Neaton, Prof., Study Chair — INSIGHT Statistical and Data Management Center, University of Minnesota
Locations (107):
- United States (76):
  - Banner University Medical Center Tucson (Site 206-004), 1625 N. Campbell Avenue, Tucson, Arizona
  - Southern Arizona VA Healthcare System (Site 074-009), 3601 S. 6th Ave., Tucson, Arizona
  - Community Regional Medical Center (Site 203-005), 2823 Fresno Street, Fresno, California
  - VA Loma Linda Healthcare System (Site 074-017), 11201 Benton Street, Loma Linda, California
  - VA Long Beach Healthcare System (Site 074-026), 5901 East 7th Street (09/151-M2), Long Beach, California
  - Keck Hospital of USC (Site 301-020), 1500 San Pablo Street, Los Angeles, California
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Blvd., Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), 757 Westwood Plaza, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian (Site 080-026), One Hoag Drive, Newport Beach, California
  - UCSF Medical Center at Mount Zion (Site 203-007), 1600 Divisadero St., San Francisco, California
  - San Francisco VAMC (Site 074-002), 4150 Clement St., San Francisco, California
  - UCSF Medical Center (Site 203-001), Moffitt-Long Hospital, 505 Parnassus Ave., San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), 300 Pasteur Dr., Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Site 066-002), 1124 W. Carson Street, CDCRC Building, Torrance, California
  - University of Colorado Hospital (Site 204-001), 12605 E. 16th Avenue, Aurora, Colorado
  - Denver Public Health (Site 017-004), 660 Bannock St., MC2600 (Infectious Disease Clinic), Denver, Colorado
  - National Jewish Health / St. Joseph Hospital (Site 204-003), 1400 Jackson Street, Denver, Colorado
  - MedStar Georgetown University Hospital (Site 067-001), 3800 Reservoir Road NW, Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), 50 Irving Street NW, Washington D.C., District of Columbia
  - Bay Pines VAMC (Site 074-004), 10000 Bay Pines Blvd., Bldg. 100, Room 5B-104, Bay Pines, Florida
  - Baycare Health System (Site 301-025), Morton Plant Hospital, 300 Pinellas Street, Clearwater, Florida
  - North Florida/South Georgia Veterans Health System (Site 074-011), 1601 SW. Archer Road, Gainesville, Florida
  - Memorial Healthcare System (Site 648-002), Memorial Regional Hospital, 3501 Johnson Street, Hollywood, Florida
  - Miami VAMC (Site 074-003), 1201 NW 16 Street, Miami, Florida
  - Hillsborough County Health Department, University of South Florida (Site 032-001), Tampa, Florida
  - Emory University (Site 301-008), The Emory Clinic, Bldg. A, Suite 2236, 1365 Clifton Rd., NE, Atlanta, Georgia
  - Lutheran Medical Group (Site 301-010), 7916 W. Jefferson Boulevard, Fort Wayne, Indiana
  - Cotton O'Neil Clinical Research Center (Site 080-030), Stormont Vail Health, 1500 SW 10th Avenue, Topeka, Kansas
  - University of Kentucky Hospital (Site 210-004), 1000 South Limestone St., Lexington, Kentucky
  - Ochsner Clinic Foundation (Site 301-015), 1514 Jefferson Highway, New Orleans, Louisiana
  - University of Maryland Medical Center (Site 301-019), 22 South Greene Street, Baltimore, Maryland
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Site 202-001), 330 Brookline Ave., Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), 759 Chestnut Street, Springfield, Massachusetts
  - University of Michigan (Site 205-001), 1500 East Medical Center Drive, Ann Arbor, Michigan
  - Henry Ford Health System, Henry Ford Hospital (Site 014-001), 2799 W. Grand Blvd., Detroit, Michigan
  - Minneapolis Heart Institute Foundation (Site 301-026), Abbott Northwestern Hospital, 920 E 28th St. #100, Minneapolis, Minnesota
  - Hennepin Healthcare (Site 027-001), 701 Park Avenue, Minneapolis, Minnesota
  - Minneapolis VA Health Care System (Site 105-001), 1 Veterans Drive, Bldg 70, Minneapolis, Minnesota
  - University of Mississippi Medical Center (Site 202-005), 2500 North State Street, Jackson, Mississippi
  - VA St. Louis Healthcare System (Site 074-027), 915 North Grand Blvd., Rm. C201, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital (Site 301-024), One Medical Center Drive, Lebanon, New Hampshire
  - Cooper University Hospital (Site 019-001), One Cooper Plaza, Camden, New Jersey
  - Ichan School of Medicine at Mount Sinai (Site 301-012), One Gustave L. Levy Place, Box 1620, New York, New York
  - Lincoln Medical Center (New York Health and Hospitals/Lincoln) (Site 003-016), 234 E. 149th Street, The Bronx, New York
  - Montefiore Medical Center Weiler Hospital (Site 206-003), 1825 Eastchester Road, The Bronx, New York
  - Montefiore Medical Center Moses Hospital (Site 206-001), 111 E. 210th Street, The Bronx, New York
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest University Health Sciences (Site 210-001), Medical Center Blvd, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (Site 207-003), 234 Goodman Ave., Cincinnati, Ohio
  - Cleveland Clinic Fairview Hospital (Site 207-005), 18101 Lorain Avenue, Cleveland, Ohio
  - Cleveland Clinic Foundation (Site 207-001), 9500 Euclid Avenue, Cleveland, Ohio
  - Cleveland Clinic Marymount Hospital (Site 207-006), 12300 McCraken Road, Garfield Heights, Ohio
  - Oregon Health & Science University (Site 208-003), 3181 SW Sam Jackson Park Rd., Portland, Oregon
  - UPMC Magee-Womens Hospital (Site 209-003), 300 Halket Street, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital (Site 209-001), 200 Lothrop Street, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital (Site 209-005), 5230 Centre Avenue, Pittsburgh, Pennsylvania
  - Rhode Island Hospital (Site 080-036), 593 Eddy Street, Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), 164 Summit Ave., Providence, Rhode Island
  - MUSC Research Nexus Clinic (Site 210-002), 96 Jonathan Lucas St., CSB 214, Charleston, South Carolina
  - VA TVHS Nashville Campus (Site 074-022), 1310 24th Avenue South, Nashville, Tennessee
  - Vanderbilt University Medical Center (Site 212-001), 1211 Medical Center Drive, Nashville, Tennessee
  - CHRISTUS Spohn Shoreline Hospital (Site 080-001), 600 Elizabeth Street, Corpus Christi, Texas
  - Parkland Health and Hospital Systems (Site 084-002), 5200 Harry Hines Blvd, Dallas, Texas
  - UT Southwestern Medical Center (Site 084-001), 1936 Amelia Court, 2nd Floor, Dallas, Texas
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center (MEDV AMC) (Site 074-006), 2002 Holcombe Blvd., Houston, Texas
  - Texas Heart Institute (Site 301-017), 6770 Bertner, MC4-266, Houston, Texas
  - CHRISTUS Good Shepherd Medical Center (Site 080-031), 700 E. Marshall Ave., Longview, Texas
  - Intermountain Medical Center (Site 211-001), 5121 South Cottonwood Street, Murray, Utah
  - University of Utah Hospital (Site 211-002), 419 Wakara Way, Suite 207, Salt Lake City, Utah
  - LDS Hospital (Site 211-004), 8th Ave. C Street, Salt Lake City, Utah
  - University of Virginia Health Systems (Site 301-021), 1215 Lee Street, Charlottesville, Virginia
  - Salem VA Medical Center (Site 074-014), 1970 Roanoke Blvd., Salem, Virginia
  - Swedish Hospital First Hill (Site 208-005), 747 Broadway, Seattle, Washington
  - West Virginia University (Site 301-023), One Medical Center Drive, Morgantown, West Virginia
- Denmark (10):
  - Aalborg Hospital (Site 625-005), Hobrovej 18, Aalborg
  - Aarhus Universitetshospital, Skejby (Site 625-002), Department of Infectious Diseases, Palle Juul-Hensens Boulevard 99, Aarhus N
  - Bispebjerg Hospital (Site 625-013), Bispebjerg Bakke 23, Copenhagen
  - Righospitalet (Site 625-006), Blegdamsvej 9,, Copenhagen Ø
  - Herlev/Gentofte Hospital (Site 625-012), Medicinsk Afdeling, Herlev Ringvej 75, Herlev
  - Nordsjællands Hospital (Site 625-009), Dyrehavevej 29, Hillerød
  - Hvidovre University Hospital, Department of Infectious Diseases (Site 625-001), Kettegård allé 30, Hvidovre
  - Kolding Sygehus (Site 625-011), Medicinsk Afdeling, Sygehusvej 24, Kolding
  - Odense University Hospital (Site 625-004), Infektionsmedicinsk Forskningsenhed, J.B. Winsløwsgade 4, Odense
  - Zealand University Hospital, Roskilde (Site 625-010), Sygehusvej 10, Roskilde
- Wojewódzki Szpital Zakazny (Site 625-302), Wolska 37, Warsaw, Poland
- Tan Tock Seng Hospital (Site 612-201), National Centre for Infectious Diseases (NCID), 11 Jalan Tan Tock Seng, Singapore, Singapore
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol (Site 626-003), Infectious Disease Unit, Second Floor, Building Maternal, Road Canyet s/n, Badalona, Barcelona
  - Hospital Universitari Arnau de Vilanova (Site 626-035), Av. Alcalde Rovira Roure 80, Lleida, Leida
  - Hospital Del Mar (Site 626-025), Paseo Maritimo 25-29, Barcelona
  - Hospital Universitari Vall d'Hebron (Site 626-033), Passeig de la Vall d'Hebron 119-129, Barcelona
  - Hospital Clínic de Barcelona (Site 626-004), Carrer de Villaroel 170, Barcelona
  - Hospital Universitario de Bellvitge (Site 626-034), Carrer de la Feixa Llarga, s/n, Barcelona
  - Hospital General Universitario Gregorio Marañón (Site 626-001), Dr. Esquerdo, 46, Madrid
  - Hospital Clínico San Carlos (Site 626-017), Enfermedades infecciosas, C/Martin Lagos CN, Madrid
  - UCICEC (Clinical Trial Unit) Hospital Universitario La Paz (Site 626-012), Paseo de la Castellana 261, 2a planta Hospital Maternal, Madrid
- University Hospital Zurich (Site 621-201), Department of Infectious Diseases and Hospital Epidemiology, Raemistrasse 100, Zurich, Canton of Zurich, Switzerland
- Uganda (6):
  - MRC/UVRI and LSHTM Uganda Research Unit (Site 634-601), Entebbe Regional Referral Hospital, Entebbe
  - Gulu Regional Referral Hospital (Site 634-603), Laroo Division, PO Box 160, Gulu
  - Makerere University Lung Institute (Site 634-604), New Mulago Hospital Complex, Mulago Hill, Kampala
  - St. Francis Hospital, Nsambya (Site 634-607), Nsambya Road Nsambya Hill, P.O. Box 7146, Kampala
  - Lira Regional Referral Hospital (Site 634-605), Lira
  - Masaka Regional Referral Hospital (Site 634-606), MRC/UVRI and LSHTM Uganda Research Unit, Plot 6 Circle Road, PO Box 556, Masaka
- United Kingdom (3):
  - Royal Victoria Infirmary (Site 634-007), Queen Victoria Road, Newcastle upon Tyne, Northumbria
  - Royal Free Hospital (Site 634-006), Pond Street, Hampstead, London
  - Guy's and St. Thomas' NHS Foundation Trust (Site 634-011), London

REFERENCES:
- [Result] ACTIV-3/Therapeutics for Inpatients with COVID-19 (TICO) Study Group. Efficacy and safety of two neutralising monoclonal antibody therapies, sotrovimab and BRII-196 plus BRII-198, for adults hospitalised with COVID-19 (TICO): a randomised controlled trial. Lancet Infect Dis. 2022 May;22(5):622-635. doi: 10.1016/S1473-3099(21)00751-9. Epub 2021 Dec 23. PMID 34953520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 43 sites in 4 countries (Denmark, Switzerland, Poland, USA). The first subject was enrolled on 16 Dec 2020 and the last subject was enrolled on 1 Mar 2021.
Groups:
- BRII-196/BRII-198 Plus SOC: * BRII-196 1000 mg solution; administered as IV infusion
  * BRII-198 1000 mg solution; administered as IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  BRII-196: BRII-196 is a fully human immunoglobulin G (IgG)-1 monoclonal antibody (mAb) derived from antibody P2C-1F11 that was isolated directly from human B cells of a convalescent COVID-19 patient.
  BRII-198: BRII-198 is a fully human immunoglobulin G (IgG)-1 monoclonal antibody (mAb) derived from antibody P2B-1G5 that was isolated directly from human B cells of a convalescent COVID-19 patient.
  Remdesivir: Antiviral agent
- Placebo Plus SOC: * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Placebo: Commercially available 0.9% sodium chloride solution
  Remdesivir: Antiviral agent
Period: Overall Study
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
Started | 176 | 177
Completed | 176 | 177
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC | Total
Number analyzed (Participants) | 176 | 177 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (14.4) | 59.5 (14.8) | 59.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 74 | 152
  Male | 98 | 103 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 32 | 66
  Not Hispanic or Latino | 142 | 145 | 287
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12 | 9 | 21
  American Indian or Alaska Native | 0 | 2 | 2
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Black or African American | 37 | 37 | 74
  White | 105 | 108 | 213
  More than one race | 1 | 0 | 1
  Other | 8 | 5 | 13
  Only ethnicity reported | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Ordinal Outcome on Day 5
Description: Ordinal outcome with 7 mutually exclusive categories
Time Frame: Status on Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 173 | 177
Participants
  7 = Death | 1 | 1
  6 = Invasive ventilation, ECMO, mechanical circulatory support, new renal replacement therapy | 4 | 3
  5 = Non-invasive ventilation or high flow oxygen | 15 | 14
  4 = Supplement oxygen (≥4 L/min or ≥4 L/min above baseline, but not high flow oxygen) | 18 | 20
  3 = Supplement oxygen (<4 L/min or <4 L/min above baseline, but not high flow oxygen) | 33 | 42
  2 = Limiting symptoms due to COVID-19, but not need of new or increased oxygen from baseline | 58 | 57
  1 = No limiting symptoms due to COVID-19 | 44 | 40

2. Secondary Outcome: Number of Participants Who Died From All Causes
Description: All-cause mortality
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 176 | 177
Participants | 15 | 13

3. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 5
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 5
Time Frame: Through Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 176 | 177
Participants | 46 | 43

4. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 28
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 28
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 176 | 177
Participants | 58 | 57

5. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 90
Description: Death, SAE, clinical organ failure, serious infections through Day 90
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 176 | 177
Participants | 45 | 47

ADVERSE EVENTS:
Time Frame: 90 days
Description: Only Grade 3 or 4 AEs were collected.
Arm/Group | BRII-196/BRII-198 Plus SOC | Placebo Plus SOC
All-Cause Mortality (participants affected / at risk) | 15/176 | 13/177
Serious Adverse Events (participants affected / at risk) | 13/176 | 11/177
Other Adverse Events (participants affected / at risk) | 45/176 | 40/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRII-196/BRII-198 Plus SOC (N=176) | Placebo Plus SOC (N=177)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRII-196/BRII-198 Plus SOC (N=176) | Placebo Plus SOC (N=177)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumopericardium (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 6 (6)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Oxygen consumption increased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 13 (15)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (8)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 7 (8) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ear and Labyrinth (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Trial H3 Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT05780424/Prot_000.pdf
  • Study Protocol: Master Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT05780424/Prot_001.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT05780424/SAP_002.pdf
  • Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT05780424/ICF_003.pdf